CLINICAL TRIAL: NCT05348122
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled，Dulaglutide-controlled Phase Ⅱ Trial Exploring Optimal Dosing Regimen for TG103 Injection Monotherapy in Type 2 Diabetes
Brief Title: A Study of TG103 Injection in Type 2 Diabetes Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSA1803-008
Record Dates: First submitted 2022-04-06; First posted 2022-04-27 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- TG103, 15 mg,Q2W (Experimental): TG103 (15 mg) will be administered via subcutaneous injection once every two weeks in subjects with type 2 diabetes.
  Interventions: Drug: TG103,Q2W
- TG103, 22.5 mg,Q2W (Experimental): TG103 (22.5 mg) will be administered via subcutaneous injection once every two weeks in subjects with type 2 diabetes.
  Interventions: Drug: TG103,Q2W
- Placebo,Q2W (Placebo Comparator): Placebo will be administered via subcutaneous injection once every two weeks in subjects with type 2 diabetes.
  Interventions: Drug: Placebo,Q2W
- TG103, 7.5 mg,QW (Experimental): TG103 (7.5 mg) will be administered via subcutaneous injection once weekly in subjects with type 2 diabetes.
  Interventions: Drug: TG103,QW
- TG103, 15 mg,QW (Experimental): TG103 (15 mg) will be administered via subcutaneous injection once weekly in subjects with type 2 diabetes.
  Interventions: Drug: TG103,QW
- Placebo,QW (Placebo Comparator): Placebo will be administered via subcutaneous injection once weekly in subjects with type 2 diabetes.
  Interventions: Drug: Placebo,QW
- Dulaglutide,QW (Active Comparator): Dulaglutide will be administered via subcutaneous injection once weekly in subjects with type 2 diabetes.
  Interventions: Drug: Dulaglutide,QW

INTERVENTIONS:
Drug: TG103,Q2W — TG103 injection will be administered via subcutaneous injection once every two weeks in subjects with type 2 diabetes.
  Other Names: TG103 injection, subcutaneous injection,Q2W
  Arms: TG103, 15 mg,Q2W; TG103, 22.5 mg,Q2W
Drug: TG103,QW — TG103 injection will be administered via subcutaneous injection once weekly in subjects with type 2 diabetes.
  Other Names: TG103 injection, subcutaneous injection,QW
  Arms: TG103, 15 mg,QW; TG103, 7.5 mg,QW
Drug: Placebo,Q2W — Placebo will be administered via subcutaneous injection once every two weeks in subjects with type 2 diabetes.
  Other Names: Placebo, subcutaneous injection,Q2W
  Arms: Placebo,Q2W
Drug: Placebo,QW — Placebo will be administered via subcutaneous injection once weekly in subjects with type 2 diabetes.
  Other Names: Placebo, subcutaneous injection,QW
  Arms: Placebo,QW
Drug: Dulaglutide,QW — Dulaglutide will be administered via subcutaneous injection once weekly in subjects with type 2 diabetes.
  Other Names: Dulaglutide,subcutaneous injection,QW
  Arms: Dulaglutide,QW

SUMMARY:
The primary objective of this trial is to evaluate the efficacy of different doses and frequencies of administration of TG103 injection in the treatment of type 2 diabetes.

DETAILED DESCRIPTION:
This trial is a randomized, double-blind, placebo-parallel, Dulaglutide-controlled，multicenter phase Ⅱ clinical trial. The whole trial consists of two parts, Part A and Part B, and 240 subjects are planned to be enrolled. Part A will be divided into three groups: TG103 15 mg group, TG103 22.5 mg group and placebo group, given once every two weeks (Q2W); Part B will be divided into four groups: TG103 7.5mg dose group, TG103 15 mg dose group ,placebo group and Dulaglutide group, once a week (QW). After Part A enrollment is completed, Part B will continue to be enrolled. The trial will include a screening period of up to 2 weeks, an initiation period of 2 weeks, a double-blind treatment period of 16 weeks, and a safety follow-up period of 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes ;
* Aged 18 to 75 years (inclusive), no gender limitation;
* Body Mass Index (BMI): 18.5≤BMI≤40;
* Poor blood glucose control after diet and exercise alone without hypoglycemic drug treatment. Not treated with hypoglycemic drugs is defined as:Have not received hypoglycemic drugs before screening, or have received hypoglycemic drugs before screening, but have not received hypoglycemic drugs within 8 weeks before screening; and continuous use of insulin for no more than 14 days (except gestational diabetes) and/or the continuous use of another hypoglycemic drug for no more than 4 weeks within 1 year prior to screening;
* HbA1c must meet the following criteria:Screening: 7.5% ≤ HbA1c ≤ 11.0% (Local laboratory);Baseline: 7.0% ≤ HbA1c ≤ 10.5% (Central laboratory)
* Subjects of childbearing potential must use reliable methods of contraception throughout the study period and at least 3 months after the last dose to avoid pregnancy in female subjects or pregnancy in the male subject's partner;
* Must be able to accurately use home glucose meter for self-glucose monitoring;
* Be able to understand and follow the trial procedure, voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

* Type 1 diabetes;
* Body weight change more than 5% within 1 month prior to screening;
* Receive any of the following medications:Prior discontinuation of DPP-4 inhibitors or GLP-1 receptor agonists for efficacy, tolerability, and safety reasons;Systemic glucocorticoid and growth hormone have been used within 8 weeks before screening or before randomization;
* History of grade 3 hypoglycemia ≥2 times within 6 months prior to screening, or grade 3 hypoglycemia prior to screening to randomization;
* Acute complications of diabetes, such as diabetic ketoacidosis and hyperglycemia, occurred ≥1 time within 6 months prior to screening, or prior to randomization;
* Severe chronic complications of diabetes (e.g., proliferative diabetic retinopathy, severe diabetic neuropathy, diabetic foot, etc.) within 6 months prior to screening
* History of acute or chronic pancreatitis prior to screening, or acute or chronic pancreatitis prior to randomization;
* Subjects with clinically significant gastric emptying abnormalities (e.g., gastric outlet obstruction), severe chronic gastrointestinal diseases (e.g., gastroparesis, inflammatory bowel disease, or intestinal obstruction) within 6 months prior to screening, or prior to randomization, long-term use of drugs that directly affect gastrointestinal motility, or gastrointestinal surgery that affects gastric emptying;
* Any of the following cardiovascular events within 6 months prior to screening, or prior to randomization: unstable angina pectoris, myocardial infarction, coronary artery bypass grafting, coronary stent implantation, moderate or severe congestive heart failure (NYHA grade III or IV), atrial or ventricular arrhythmia (e.g., atrial fibrillation, ventricular tachycardia, etc.), pacemaker or defibrillator implantation; Or subjects with Ⅱ or Ⅲ degree atrioventricular block, long QT syndrome or prolonged QTcF interval (QTcF: male >450 ms, female >470 ms) on 12-lead ECG, or signs of heart disease with significant clinical symptoms at screening;
* Hemorrhagic stroke or acute ischemic stroke disease occurred within 6 months prior to screening, or prior to randomization;
* Having a history of serious respiratory tract, central nervous system (such as epilepsy, etc.) and psychiatric diseases (such as depression, anxiety, etc.) during screening; Or have a history of other diseases that may endanger the safety of the subject and that the investigator deems inappropriate for enrollment;
* Any type of malignant tumor treated or untreated within 5 years prior to screening or prior to randomization (except clinically cured basal cell carcinoma or carcinoma in situ);
* Severe or acute infection within 4 weeks prior to screening, or refractory urinary tract or genital infection within 6 months prior to screening;
* Having a significant blood system disease (e.g., aplastic anemia, myelodysplastic syndrome) or any disease causing hemolysis or red blood cell instability (e.g., malaria) at screening or prior to randomization;
* Subjects with thyroid dysfunction that cannot be controlled by a stable drug dose at screening, or with clinically significant abnormalities in thyroid function examination results requiring drug treatment at screening ;
* Personal or family history of medullary thyroid cancer (MTC) or type 2 multiple endocrine tumor syndrome at screening;
* Systolic blood pressure ≥ 160mmHg or diastolic blood pressure ≥ 100mmHg at screening or before randomization;
* Any of the following abnormalities during screening or prior to randomization of laboratory tests:FPG≥13.9 mmol/L;ALT or AST≥2.5×ULN;Total bilirubin (TBiL) ≥1.5×ULN;Triglyceride >5.7 mmol/L;eGFR<60 mL/(min*1.73 m^2);Serum amylase and/or lipase ≥3×ULN (if lipase cannot be detected in some centers, amylase alone is acceptable);Hemoglobin <100 g/L;Calcitonin≥50 ng/L(pg/mL);
* Serological examination:Human immunodeficiency virus antibody or treponema pallidum antibody is positive;Hepatitis C antibody is positive;Hepatitis B surface antigen is positive, and the quantitative detection result of HBV DNA was higher than the lower limit of the detection reference range;
* Known allergy to the test drug, Empagliflozin , or related excipients;
* Subjects who underwent major surgery within 3 months prior to screening, or who lost more than 400 mL blood due to blood donation or other reasons within 3 months prior to screening;
* Average alcohol intake more than 21 units of alcohol (male)/14 units of alcohol (female) per week within the 3 months prior to screening (1 unit ≈360 mL beer, or 45 mL spirits with 40% alcohol content, or 150 mL wine);
* Subject participated in any drug or medical device clinical study within 3 months prior to screening (except for screening failure);
* Pregnant or lactating female;
* Not suitable for this study in the investigator's opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in glycosylated hemoglobin (HbA1c) from baseline to week 17 | Baseline through Day 113
  Changes in glycosylated hemoglobin (HbA1c) from baseline to week 17

SECONDARY OUTCOMES:
Changes in glycosylated hemoglobin (HbA1c) from baseline to week 9 | Baseline through Day57
  Changes in glycosylated hemoglobin (HbA1c) from baseline to week 9
The percentage of HbA1c≤6.5% and the percentage of HbA1c≤7% at week 9 and 17 | Day57 and 113
  The percentage of HbA1c≤6.5% and the percentage of HbA1c≤7% at week 9 and 17
Change in fasting plasma glucose (FPG) from baseline to week 9 and 17 | Baseline through Day57 and 113
  Change in fasting plasma glucose (FPG) from baseline to week 9 and 17
Change in weight from baseline to week 9 and 17 | Baseline through Day57 and 113
  Change in weight from baseline to week 9 and 17
Mean postprandial blood glucose increment and change in mean postprandial blood glucose from baseline at 7-point Self-monitored Blood Glucose (SMBG) Profile. | Baseline through Day113
  Mean postprandial blood glucose increment and change in mean postprandial blood glucose from baseline at 7-point Self-monitored Blood Glucose (SMBG) Profile.
Change in 7-point Self-monitored Blood Glucose (SMBG) Profile. | Baseline through Day113
  Change in 7-point Self-monitored Blood Glucose (SMBG) Profile.
Change in blood lipids (triglycerides, total cholesterol, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol) from baseline to week 17. | Baseline through Day113
  Change in blood lipids (triglycerides, total cholesterol, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol) from baseline to week 17.
Proportion of subjects receiving remedial therapy at week 17 | Day113
  Proportion of subjects receiving remedial therapy at week 17
Number of TEAEs and SAEs from baseline to week 17 | Day-14 through Day 113
  Number of TEAEs and SAEs from baseline to week 17
Ctrough will be measured once every 4 week until week 17 | Day1, 29, 57, 85 and 113
  Ctrough will be measured once every 4 week until week 17
The occurrence of TG103 anti-drug antibodies (ADA) and neutralizing antibody (Nab). | Day1, 29, 57, 85, 113 and127
  The occurrence of TG103 anti-drug antibodies (ADA) and neutralizing antibody (Nab).

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, Principal Investigator — Peking University People's Hospital
Locations (1):
- Gao Huanhuan, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No